CLINICAL TRIAL: NCT01797536
Title: A Three-Part, Open-Label, Single-Dose Study to Investigate the Influence of Hepatic Insufficiency on the Pharmacokinetics of MK-8742
Brief Title: The Influence of Hepatic Insufficiency on the Pharmacokinetics of Elbasvir (MK-8742) (MK-8742-009)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Celerion (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8742-009
Record Dates: First submitted 2013-02-20; First posted 2013-02-22 (Estimated); Results first posted 2016-11-18 (Estimated); Last update posted 2018-10-25 (Actual); Status verified 2018-09

CONDITIONS: Hepatic Insufficiency
MeSH Terms: conditions — Hepatic Insufficiency | interventions — elbasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Mild Hepatic Insufficiency (Experimental): Single oral dose of 5 x 10 mg capsules of elbasvir administered to participants with mild hepatic insufficiency, defined as a score of 5 to 6 on the Child-Pugh scale
  Interventions: Drug: Elbasvir
- Moderate Hepatic Insufficiency (Experimental): Single oral dose of 5 x 10 mg capsules of elbasvir administered to participants with moderate hepatic insufficiency, defined as a score of 7 to 9 on the Child-Pugh scale
  Interventions: Drug: Elbasvir
- Severe Hepatic Insufficiency (Experimental): Single oral dose of 5 x 10 mg capsules of elbasvir administered to participants with severe hepatic insufficiency, defined as a score of 10 to 15 on the Child-Pugh scale
  Interventions: Drug: Elbasvir
- Healthy Participants (Experimental): Single oral dose of 5 x 10 mg capsules of elbasvir administered to participants matched to the mean of all hepatic insufficiency participants for age, gender, and weight
  Interventions: Drug: Elbasvir

INTERVENTIONS:
Drug: Elbasvir

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics (PK) profile of elbasvir (MK-8742) after a single dose to participants with mild, moderate, or severe hepatic insufficiency compared with healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) 19 - 40 kg/m^2, inclusive
* In good health based on medical history, physical examination, vital signs, and laboratory safety tests
* No clinically significant abnormality on electrocardiogram (ECG)
* For participants with hepatic insufficiency only, diagnosis of chronic (> 6 months), stable (no acute episodes of illness within the previous 2 months due to deterioration in hepatic function) hepatic insufficiency with features of cirrhosis due to any cause
* For participants with hepatic insufficiency only, score on the Child-Pugh scale must range from 5 to 6 for mild hepatic insufficiency, from 7 to 9 for moderate hepatic insufficiency, and from 10 to 15 for severe hepatic insufficiency
* Females of childbearing potential must be either be sexually inactive (abstinent) for 14 days before study drug administration and throughout the study or be using an acceptable method of birth control
* Females of non-childbearing potential must have undergone sterilization procedures at least 6 months before Study Day 1
* Non-vasectomized males must agree to use a condom with spermicide or abstain from sexual intercourse during the study and for 3 months after study drug administration
* Ability to swallow multiple capsules

Exclusion Criteria:

* Previously enrolled in this study
* Mentally or legally incapacitated, significant emotional problems at the time of screening or expected during the conduct of the study, or a history of a clinically significant psychiatric disorder over the last 5 years
* History or presence of significant cardiovascular, pulmonary, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurological disease
* History of any illness that might confound the results of the study or pose an additional risk to the participant by participating in the study
* For participants with hepatic insufficiency only, estimated creatinine clearance (CrCl) ≤30 mL/min based on the Cockcroft-Gault equation at screening
* History or presence of drug abuse within the past 2 years
* For healthy participants only, history of alcoholism within the past 2 years
* Females who are pregnant or lactating
* Positive results for the urine drug screen at screening or check-in
* Positive results at screening or history of human immunodeficiency virus (HIV) or untreated hepatitis C virus (HCV); HCV ribonucleic acid (RNA)-negative participants documented to be cured following anti-HCV treatment are eligible
* For healthy participants only, positive results at screening for hepatitis B surface antigen (HBsAg)
* Use of any drugs or substances known to be strong inhibitors of cytochrome P450 3A4 (CYP3A4) enzymes and/or P-glycoprotein (P-gp) or any inhibitors of organic anion transporting peptide 1B (OATP1B) within 14 days or 5-times the half-life of the product (for healthy participants) or which cannot be discontinued at least 14 days or 5 times the half-life of the product (for hepatic insufficiency participants) before study drug administration and throughout the study
* Use of any drugs or substances known to be strong inducers of CYP3A4 enzymes and/or P-gp, including St-John's Wort or rifampin, within 28 days or 5 times the half-life of the product before study drug administration
* Currently use of any medication or substance which cannot be discontinued or maintained at a steady dose and regimen at least 14 days before study drug administration and throughout the study
* For healthy participants only, on a special diet within 28 days before study drug administration
* Blood donation >500 mL or significant blood loss within 56 days before study drug administration
* Plasma donation within 7 days before study drug administration
* Participation in another clinical study within 28 days before study drug administration

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-03-06 (Actual); Primary Completion 2014-08-20 (Actual); Study Completion 2014-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (2):
- United States (2):
  - Call for Information (Investigational Site 0003), Miami, Florida
  - Call for Information (Investigational Site 0001), Orlando, Florida

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Marshall WL, Feng HP, Wenning L, Garrett G, Huang X, Liu F, Panebianco D, Caro L, Fandozzi C, Lasseter KC, Preston RA, Marbury T, Butterton JR, Iwamoto M, Yeh WW. Pharmacokinetics, Safety, and Tolerability of Single-Dose Elbasvir in Participants with Hepatic Impairment. Eur J Drug Metab Pharmacokinet. 2018 Jun;43(3):321-329. doi: 10.1007/s13318-017-0451-9. PMID 29247332

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 3 participants from the mild insufficiency arm were mistakenly reenrolled into the moderate arm and received a 2nd single dose of study drug. Data for these 3 participants were excluded from pharmacokinetic analysis of the moderate arm but were included in the safety analysis. An additional 3 participants were enrolled in the moderate arm.
Period: Overall Study
Arm/Group | Mild Hepatic Insufficiency | Moderate Hepatic Insufficiency | Severe Hepatic Insufficiency | Healthy Participants
Started | 8 | 11 (Includes 3 participants from mild arm who were mistakenly re-enrolled and also dosed in moderate arm) | 7 | 8
Completed | 8 | 10 | 7 | 8
Not Completed | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mild Hepatic Insufficiency | Moderate Hepatic Insufficiency | Severe Hepatic Insufficiency | Healthy Participants | Total
Number analyzed (Participants) | 8 | 11 | 7 | 8 | 34
Age, Continuous [Mean (Full Range); unit: Years] | 54 [39 to 66] | 54 [42 to 68] | 56 [48 to 62] | 54 [46 to 69] | 54.35 [39 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 4 | 2 | 7
  Male | 8 | 10 | 3 | 6 | 27

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve From 0 to Infinity (AUC0-inf) of Elbasvir
Description: Blood samples were collected at predose and Hours 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 48, 96, 144, and 168 to determine the AUC0-inf of elbasvir.
Time Frame: Predose and Hours 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 48, 96, 144, and 168
Population: Participants who complied with the protocol sufficiently to ensure that generated data were likely to exhibit the effects of treatment and had available data for the endpoint. Moderate arm summary excludes data for 3 participants incorrectly re-enrolled and dosed in moderate arm after completing dosing and follow-up in the mild insufficiency arm.
Measure: Geometric Mean (95% Confidence Interval); unit: μM•hr
Arm/Group | Mild Hepatic Insufficiency | Moderate Hepatic Insufficiency | Severe Hepatic Insufficiency | Healthy Participants
Number analyzed (Participants) | 8 | 7 | 7 | 8
μM•hr | 1.56 [0.95 to 2.57] | 1.86 [1.10 to 3.16] | 2.28 [1.34 to 3.87] | 2.58 [1.58 to 4.24]
Statistical Analysis 1: Comparison: Mild Hepatic Insufficiency vs Healthy Participants; Back-transformed least-squares mean and confidence interval from linear fixed effect model performed on natural log-transformed values; Test type: Superiority or Other; Geometric Mean Ratio (GMR) = 0.61, 90% CI 2-sided [0.34 to 1.08] — GMR= Mild Hepatic Insufficiency Geometric Mean (GM) divided by Healthy Control GM
Statistical Analysis 2: Comparison: Moderate Hepatic Insufficiency vs Healthy Participants; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; GMR = 0.72, 90% CI 2-sided [0.40 to 1.31] — GMR = Moderate Hepatic Insufficiency GM divided by Healthy Control GM
Statistical Analysis 3: Comparison: Severe Hepatic Insufficiency vs Healthy Participants; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; GMR = 0.88, 90% CI 2-sided [0.48 to 1.61] — GMR = Severe Hepatic Insufficiency GM divided by Healthy Control GM

2. Primary Outcome: Area Under the Curve From 0 to 24 Hours (AUC0-24hr) of Elbasvir
Description: Blood samples were collected at predose and Hours 0.5, 1, 2, 3, 4, 6, 8, 12, 16, and 24 to determine the AUC0-24hr of elbasvir.
Time Frame: Predose and Hours 0.5, 1, 2, 3, 4, , 6, 8, 12, 16, and 24
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: μM•hr
Arm/Group | Mild Hepatic Insufficiency | Moderate Hepatic Insufficiency | Severe Hepatic Insufficiency | Healthy Participants
Number analyzed (Participants) | 8 | 7 | 7 | 8
μM•hr | 0.87 [0.54 to 1.41] | 0.92 [0.55 to 1.55] | 0.92 [0.55 to 1.54] | 1.45 [0.90 to 2.35]
Statistical Analysis 1: Comparison: Mild Hepatic Insufficiency vs Healthy Participants; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; GMR = 0.60, 90% CI 2-sided [0.34 to 1.05] — GMR = Mild Hepatic Insufficiency GM divided by Healthy Control GM
Statistical Analysis 2: Comparison: Moderate Hepatic Insufficiency vs Healthy Participants; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; GMR = 0.64, 90% CI 2-sided [0.35 to 1.14] — GMR = Moderate Hepatic Insufficiency GM divided by Healthy Control GM
Statistical Analysis 3: Comparison: Severe Hepatic Insufficiency vs Healthy Participants; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; GMR = 0.63, 90% CI 2-sided [0.35 to 1.13] — GMR = Severe Hepatic Insufficiency GM divided by Healthy Control GM

3. Primary Outcome: Maximum Concentration (Cmax) of Elbasvir
Description: Blood samples were collected at predose and Hours 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 48, 96, 144, and 168 to determine the Cmax of Elbasvir.
Time Frame: Predose and Hours 0.5, 1, 2, 3, 4, , 6, 8, 12, 16, 24, 48, 96, 144, and 168
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: nM
Arm/Group | Mild Hepatic Insufficiency | Moderate Hepatic Insufficiency | Severe Hepatic Insufficiency | Healthy Participants
Number analyzed (Participants) | 8 | 8 | 7 | 8
nM | 70.1 [42.3 to 116.0] | 83.0 [50.1 to 137.0] | 70.7 [41.3 to 121.0] | 121.0 [73.1 to 200.0]
Statistical Analysis 1: Comparison: Mild Hepatic Insufficiency vs Healthy Participants; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; GMR = 0.58, 90% CI 2-sided [0.32 to 1.05] — GMR = Mild Hepatic Insufficiency GM divided by Healthy Control GM
Statistical Analysis 2: Comparison: Moderate Hepatic Insufficiency vs Healthy Participants; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; GMR = 0.64, 90% CI 2-sided [0.35 to 1.14] — GMR = Moderate Hepatic Insufficiency GM divided by Healthy Control GM
Statistical Analysis 3: Comparison: Severe Hepatic Insufficiency vs Healthy Participants; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; GMR = 0.58, 90% CI 2-sided [0.32 to 1.08] — GMR = Severe Hepatic Insufficiency GM divided by Healthy Control GM

4. Primary Outcome: Concentration at 24 Hours (C24) After Dosing Elbasvir
Description: Blood samples were collected at predose and Hours 0.5, 1, 2, 3, 4, 6, 8, 12, 16, and 24, to determine the concentration of elbasvir at Hour 24 was determined.
Time Frame: Hour 24
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: nM
Arm/Group | Mild Hepatic Insufficiency | Moderate Hepatic Insufficiency | Severe Hepatic Insufficiency | Healthy Participants
Number analyzed (Participants) | 8 | 7 | 7 | 8
nM | 22.9 [14.0 to 37.5] | 25.9 [15.3 to 43.9] | 29.6 [17.4 to 50.1] | 37.7 [23.0 to 61.7]
Statistical Analysis 1: Comparison: Mild Hepatic Insufficiency vs Healthy Participants; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; GMR = 0.61, 90% CI 2-sided [0.34 to 1.08] — GMR = Mild Hepatic Insufficiency GM divided by Healthy Control GM
Statistical Analysis 2: Comparison: Moderate Hepatic Insufficiency vs Healthy Participants; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; GMR = 0.69, 90% CI 2-sided [0.38 to 1.25] — GMR = Moderate Hepatic Insufficiency GM divided by Healthy Control GM
Statistical Analysis 3: Comparison: Severe Hepatic Insufficiency vs Healthy Participants; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; GMR = 0.78, 90% CI 2-sided [0.43 to 1.43] — GMR = Severe Hepatic Insufficiency GM divided by Healthy Control GM

5. Primary Outcome: Time to Maximum Concentration (Tmax) of Elbasvir
Description: Blood samples were collected at predose and Hours 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 48, 96, 144, and 168 to determine the maximum concentration (Cmax) of elbasvir. The time to reach Cmax (Tmax) was determined.
Time Frame: Predose and Hours 0.5, 1, 2, 3, 4, , 6, 8, 12, 16, 24, 48, 96, 144, and 168
Population: as for outcome 1
Measure: Median (Full Range); unit: hour (hr)
Arm/Group | Mild Hepatic Insufficiency | Moderate Hepatic Insufficiency | Severe Hepatic Insufficiency | Healthy Participants
Number analyzed (Participants) | 8 | 8 | 7 | 8
hour (hr) | 3.50 [2.00 to 6.00] | 3.50 [2.00 to 4.00] | 4.00 [3.00 to 4.00] | 3.50 [2.00 to 4.00]

6. Primary Outcome: Apparent Terminal Half-Life (t1/2) of Elbasvir
Description: Blood samples were collected at predose and Hours 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 48, 96, 144, and 168 to determine the t1/2 of elbasvir.
Time Frame: Predose and Hours 0.5, 1, 2, 3, 4, , 6, 8, 12, 16, 24, 48, 96, 144, and 168
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | Mild Hepatic Insufficiency | Moderate Hepatic Insufficiency | Severe Hepatic Insufficiency | Healthy Participants
Number analyzed (Participants) | 8 | 7 | 7 | 8
hr | 24.80 (21.65) | 25.39 (34.24) | 33.72 (20.82) | 20.74 (12.64)

ADVERSE EVENTS:
Time Frame: up to 14 days post-dose (total of 14 days for each panel)
Description: All participants who received study medication. Includes safety data for 3 participants who were enrolled in both mild and moderate hepatic insufficiency arms and received study medication while enrolled in both arms.
Arm/Group | Mild Hepatic Insufficiency | Moderate Hepatic Insufficiency | Severe Hepatic Insufficiency | Healthy Participants
Serious Adverse Events (participants affected / at risk) | 0/8 | 1/11 | 0/7 | 0/8
Other Adverse Events (participants affected / at risk) | 1/8 | 3/11 | 0/7 | 0/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mild Hepatic Insufficiency (N=8) | Moderate Hepatic Insufficiency (N=11) | Severe Hepatic Insufficiency (N=7) | Healthy Participants (N=8)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mild Hepatic Insufficiency (N=8) | Moderate Hepatic Insufficiency (N=11) | Severe Hepatic Insufficiency (N=7) | Healthy Participants (N=8)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication timelines.